CLINICAL TRIAL: NCT06737848
Title: The Comparison of Single Catheter and Double Catheter Adrenal Vein Sampling Methods Based on the Upper Limb Approach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Army Medical University, China (Other)
Responsible Party: Principal Investigator, Li Li, Deputy Director of the department of Hypertension & Endocrinology, Daping Hospital, Army Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMCIIT241106
Record Dates: First submitted 2024-12-06; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Catheter Adrenal Vein Sampling (Experimental): Patients in the Intervention group will utilize a multifunctional catheter for bilateral adrenal vein sampling.
  Interventions: Procedure: Single catheter adrenal vein sampling
- Double Catheter Adrenal Vein Sampling (Active Comparator): Patients in this group will utilize two catheters for bilateral adrenal vein sampling.
  Interventions: Procedure: Double catheters adrenal vein sampling

INTERVENTIONS:
Procedure: Single catheter adrenal vein sampling — The clinical invasive procedure involves inserting a single catheter into the right and left adrenal veins to collect blood samples from both adrenal veins.
  Arms: Single Catheter Adrenal Vein Sampling
Procedure: Double catheters adrenal vein sampling — The clinical invasive procedure involves inserting double catheters into the right and left adrenal veins to collect blood samples from both adrenal veins.
  Arms: Double Catheter Adrenal Vein Sampling

SUMMARY:
Primary Aldosteronism (PA) is a clinical syndrome characterized by the autonomous overproduction of aldosterone by the adrenal cortex's zona glomerulosa, leading to hypertension, elevated aldosterone levels, and suppressed renin activity as the primary manifestations. Studies have shown that the prevalence of PA in an unselected hypertensive population ranges from 5% to 11% , while the prevalence in patients with resistant hypertension is approximately 20% . PA is one of the most common causes of secondary hypertension , and its prevalence increases with rising blood pressure levels. Due to the adverse effects of PA on the heart, arterial walls, and kidneys, it contributes to the occurrence of cardiovascular events, with atrial fibrillation being the most common . In summary, PA is characterized by rapid onset, significant symptoms, obscurity, and severe complications, making early diagnosis and targeted treatment essential for prevention.

This study aims to explore a quasi-selected prospective randomized controlled method to compare the clinical efficacy differences between single-catheter and dual-catheter adrenal sampling via the right upper limb approach. The study seeks to clarify the effectiveness and safety of single-catheter sampling from the upper limb, providing a more efficient and cost-effective solution for the subtype diagnosis of patients with Primary Aldosteronism (PA).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years with hypertension.
* Initial screening shows a standing aldosterone/renin ratio (ARR) > 3.7, a baseline aldosterone level > 10 ng/dl, aldosterone level > 6 ng/dl after a saline load test, or aldosterone decrease of less than 30% after a captopril suppression test, consistent with a diagnosis of primary aldosteronism.
* Voluntary participation in the trial, with signed informed consent.

Exclusion Criteria:

* Patients with an allergy to iodinated contrast agents.
* Patients who are pregnant, breastfeeding, or planning to become pregnant.
* Patients with severe comorbidities, such as renal failure, liver cirrhosis, metastatic tumors, or those who have had an acute stroke or acute myocardial infarction, as well as patients with a history of surgery within the past month.
* Patients suspected of having adrenal cortical carcinoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Success rate of left-sided adrenal vein sampling between two groups | 7 month(End of Trial)
  Biochemical analysis of puncture-point blood samples: A selection index (SI) ≥ 2, defined as the ratio of adrenal plasma cortisol concentration (PCC) to peripheral PCC, indicates successful unilateral aldosterone venous sampling (AVS).

SECONDARY OUTCOMES:
Change of material costs between two groups | 7 month(End of Trial)
Change of average operation time of left-side adrenal vein sampling between two groups | 7 month(End of Trial)
  The surgical doctor will record the operation time for adrenal vein sampling from the left adrenal vein and compare change of the average operation time between the two groups at end of the study.
Change of average fluoroscopy time of adrenal vein sampling between two groups | 7 month(End of Trial)
  Change of average fluoroscopy time of adrenal vein sampling between two groups at the end of the study.
Change of the surgical supplies cost between two groups | 7 month(End of Trial)
  Change of the surgical supplies cost between two groups at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, Study Director — Army Medical University, China

IPD SHARING:
Plan to Share IPD: No